CLINICAL TRIAL: NCT07279961
Title: A Multicenter Retrospective Study in China: the Factors Influencing the Success of Redo Surgery and Anal Function for Anastomosis Failure or Local Tumor Recurrence
Brief Title: A Multicenter Study on the Safety and Functionality Evaluation of Anastomotic Redo Surgery
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCCH-000166
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To analyze the influencing factors of the success of redo surgery due to anastomotic fistula or anastomotic recurrence after rectal cancer surgery and to evaluate the anal function of patients

DETAILED DESCRIPTION:
Redo surgery is a critical salvage strategy for anastomotic complications or local recurrence following rectal cancer resection. Despite technical feasibility, functional outcomes remain suboptimal. This study evaluated intestinal continuity restoration and anal function recovery after redo surgery, alongside prognostic factors influencing outcomes. A retrospective multicenter study analyzed 143 patients undergoing redo surgery (2015-2023) for anastomotic failure or local recurrence. Primary endpoints included anatomical restoration of intestinal continuity, while secondary endpoints assessed functional outcomes using the LARS score.

ELIGIBILITY:
Inclusion Criteria:

* Prior curative resection for primary colorectal adenocarcinoma.
* Subsequent reoperation for anastomotic failure or locoregional recurrence.
* Absence of absolute contraindications to reoperative surgery.

Exclusion Criteria:

* Primary tumors located proximal to the sigmoid colon.
* Radiologically confirmed distant metastases.
* Presence of a permanent stoma at the time of questionnaire administration.
* Insufficient literacy or cognitive function to complete study-related -questionnaires.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective, multicenter study analyzed data from a prospectively maintained redo surgery registry spanning March 2015 to March 2023. Patients were recruited from Cancer Hospital Chinese Academy of Medical Sciences,Sun Yat-sen University Sixth Affiliated Hospital and Yifu Hospital Affiliated to Nanjing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Whether postoperative patients with rectal cancer can restore intestinal continuity, that is, defecate through the anus | During the follow-up period, at least two years after rectal cancer surgery

SECONDARY OUTCOMES:
Low Anterior Rectal Syndrome (LARS) Score of patients restoring intestinal continuity | During the follow-up period, at least one year has passed since the intestinal continuity was restored

IPD SHARING:
Plan to Share IPD: No